CLINICAL TRIAL: NCT00002908
Title: PHASE II CLINICAL EVALUATION OF BRYOSTATIN 1 IN PATIENTS WITH RELAPSED NON-HODGKIN'S LYMPHOMA AND CLL
Brief Title: Bryostatin 1 in Treating Patients With Relapsed Non-Hodgkin's Lymphoma or Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000065273; P30CA022453 (NIH); WSU-C-1256; WSU-D-1256; NCI-T95-0058D
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — bryostatin 1; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bryostatin 1
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of bryostatin 1 in treating patients who have relapsed non-Hodgkin's lymphoma or chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy of bryostatin 1 administered as a 72-hour infusion in patients with relapsed non-Hodgkin's lymphoma and chronic lymphocytic leukemia. II. Gain information regarding the toxicity and tolerability of escalated vincristine doses given after each bryostatin 1 infusion in cohorts of patients who fail to respond to bryostatin alone. III. Determine the qualitative and quantitative toxic effects of bryostatin 1 in these patients. IV. Determine the duration of response and survival following treatment with bryostatin 1.

OUTLINE: All patients receive bryostatin 1 by 72-hour continuous infusion every 2 weeks until disease progression or until 2 courses beyond documentation of complete remission. Response is assessed after every 4 courses. Patients with disease progression who continue to meet the eligibility criteria receive vincristine within 2 hours after completion of each bryostatin 1 infusion. Groups of 3-6 patients receive escalated doses of vincristine until the maximum tolerated dose with bryostatin 1 is determined. Courses repeat every 2 weeks, as above; no individual dose escalation is allowed. No concurrent steroids are permitted. Patients are followed for survival.

PROJECTED ACCRUAL: A total of 25 evaluable patients with low-grade NHL or CLL will be entered over approximately 20 months if there are 2-4 responses in the first 15 patients. A total of 20 evaluable patients with intermediate- or high-grade NHL will be entered over approximately 2 years if there are 1 or 2 responses in the first 10 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: One of the following hematologic malignancies that has failed 1 or 2 prior front-line chemotherapy regimens and is ineligible for treatment of higher potential efficacy: Histologically confirmed chronic lymphocytic leukemia (CLL) Intermediate- or high-risk (RAI stage I-IV) disease Evidence of active disease required by at least one of the following for intermediate-risk CLL: One of the following B symptoms: Weight loss of 10% or more in previous 6 months Extreme fatigue Fever over 100 F without evidence of infection Night sweats Massive (more than 6 cm below left costal margin) or progressive splenomegaly Massive (more than 10 cm in longest diameter) or progressive lymphadenopathy Progressive lymphocytosis with more than 50% increase over 2-month period or anticipated doubling time of less than 12 months Progressive bone marrow failure as manifested by development or worsening of anemia and/or thrombocytopenia Autoimmune anemia and/or thrombocytopenia poorly responsive to corticosteroids Biopsy proven low-, intermediate-, or high-grade non-Hodgkin's lymphoma Transformed lymphoma allowed Measurable disease required Re-treatment on this study allowed if disease relapsed after a complete remission

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: At least 12 weeks Hematopoietic: ANC at least 1,500/mm3 (at least 1,000/mm3 in CLL patients with at least 30% marrow involvement) Platelets at least 100,000/mm3 (at least 50,000/mm3 in CLL patients with at least 30% marrow involvement) Hepatic: Bilirubin less than 1.5 mg/dL Transaminases less than 2.5 times normal Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: No history of impaired cardiac status, e.g.: Severe coronary artery disease Cardiomyopathy Uncontrolled congestive heart failure Arrhythmia Other: No known AIDS or HIV infection No second malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer In situ cervical cancer Not pregnant or nursing Effective contraception required of fertile patients during and for 2 months after study

PRIOR CONCURRENT THERAPY: No concurrent therapy Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since chemotherapy (8 weeks since nitrosoureas or mitomycin) and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since radiotherapy and recovered Surgery: Not specified Other: No prior bone marrow transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-12; Primary Completion 2000-02 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayad M. Al-Katib, MD, FACP, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States